CLINICAL TRIAL: NCT04000477
Title: Endocervical Curettage Performed With a Kevorkian Curette Versus Cytobrush in Patients With ASC-H, LSIL, ASCUS HPV Positive and Non-contributory Colposcopy (ZT3) Smear or Atypical Pap Smear With Positive HPV Test
Brief Title: Comparison of 2 Types of Cervical Specimens in Patients With a Pathological Screening Smear
Acronym: ENDOCOL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: default inclusion
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017_85; 2018-A03087-48 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-06-26; First posted 2019-06-27 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancer; Pathological Screening Smear
Keywords: Endocervical curettage; Kevorkian; Cytobrush; FCV
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kevorkian curette (Experimental)
  Interventions: Device: Kevorkian curette
- Cytobrush (Experimental)
  Interventions: Device: Cytobrush

INTERVENTIONS:
Device: Cytobrush — the brush would be inserted in full until the display of the brush in the endocervical canal disappears. A neck quadrant scan (= quarter turn) will be performed from front to back while simultaneously rotating the brush clockwise, for a total of 3 laps. This would represent 4 sweeps per turn, ie 12 sweeps in total
  Arms: Cytobrush
Device: Kevorkian curette — the colposcopist holds the curette horizontally and scrapes the endocervical canal all the way around. He realizes 1 small firm and linear movement by quarter turn or 4 movements to realize a complete turn. During this act, the curette must remain inside the canal, and during its extraction, care should be taken not to rotate it so as not to spill the collected tissue contained in the basket of the curette. The tissue material thus obtained must be rapidly immersed in formalin
  Arms: Kevorkian curette

SUMMARY:
The recommendations on the method and the realization of the cervico-uterine smears are clear. With regard to performing endocervical curettage, several methods are possible without precise consensus. In general, the Kevorkian curette is widely used. However, it is often reported by doctors and patients that curettage is painful. Some articles show that the cytobrush would be less painful. While keeping a percentage of correct curettage failures, it is sought to show that the cytobrush would improve the comfort of the patient during curettage.

ELIGIBILITY:
Inclusion Criteria:

* Women followed for a cervical pathology requiring endocervical curettage:
* AGC type (glandular cell atypia) with positive HPV test
* Frottis ASC-H, LSIL, ASCUS HPV + with non-contributive colposcopy (ZT3)

Exclusion Criteria:

* Pregnant woman
* Women under the age of 25 or over 65
* Stenosis of the neck complete or tight not allowing the possible insertion of a curette (inadequate size cervical orifice and material)
* Presence of a vaginal lesion on colposcopic examination

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients aged 25 to 65 years old whose screening smear returned pathologically and who are therefore followed in colposcopy
Enrollment: 3 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Percentage of sampling failures | once time, Baseline
  Unsatisfactory sampling will be defined by a specimen containing <20 endocervical cells, <3 epithelial flaps, and one specimen without stroma.

SECONDARY OUTCOMES:
Pain Assessment Using a Visual Analogue Scale (VAS) | once time, Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Jonard, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Service de gynécologie endocrinienne et médecine de la reproduction, Lille, France